CLINICAL TRIAL: NCT06859892
Title: Effect of Dexmedetomidine-esketamine Combination on Sleep Disturbances After Major Noncardiac Surgery: a Single-center, Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Dexmedetomidine-Esketamine Combination and Sleep Disturbances After Major Noncardiac Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Mo Li, Anesthesiologist, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-729
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Adults; Major Noncardiac Surgery; Dexmedetomidine; Esketamine; Postoperative Sleep Disturbances
Keywords: adults; major noncardiac surgery; dexmedetomidine; esketamine; postoperative sleep disturbances

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine-esketamine group (Experimental): Dexmedetomidine-esketamine combination is infused during general anesthesia and used as a supplement for patient-controlled intravenous analgesia after surgery.
  Interventions: Drug: Dexmedetomidine-esketamine combination
- Placebo group (Placebo Comparator): Placebo (normal saline) is infused during general anesthesia and used as a supplement for patient-controlled intravenous analgesia after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine-esketamine combination — Dexmedetomidine 0.4 μg/kg and esketamine 0.2 mg/kg is infused over 10 minutes before anesthesia induction. Dexmedetomidine 0.20 μg/kg/h and esketamine 0.10 mg/kg/h is then infused until 60 minutes before the expected end of surgery. Patient-controlled intravenous analgesia is established with 100 μg dexmedetomidine, 50 mg esketamine, and 100 μg sufentanil, diluted to 100 mL with normal saline, and programmed to deliver 2-mL boluses with a lock-out interval of 8 minutes and background infusion rate at 1 mL/h for up to 72 hours after surgery.
  Arms: Dexmedetomidine-esketamine group
Drug: Placebo — Placebo (normal saline) is administered in the same rate and volume as that in the dexmedetomidine-esketamine group. Patient-controlled intravenous analgesia is established with 100 μg sufentanil, diluted to 100 mL with normal saline, and programmed to deliver 2-mL boluses with a lock-out interval of 8 minutes and background infusion rate at 1 mL/h for up to 72 hours after surgery.
  Arms: Placebo group

SUMMARY:
Sleep disturbances are common early after major surgery, and are associated with delayed recovery. A previous study showed that dexmedetomidine-esketamine combination as a supplement to patient-controlled intravenous analgesia improved postoperative analgesia and subjective sleep quality in patients after scoliosis correction surgery. The purpose of this trial is to test the hypothesis that dexmedetomidine-esketamine combination used as a supplement during general anesthesia and postoperative intravenous analgesia may reduce sleep disturbances in adult after major noncardiac surgery.

DETAILED DESCRIPTION:
Sleep disturbances after surgery is usually manifested as sleep deprivation, altered circadian rhythm, and disturbed sleep structure. The reported incidence of sleep disturbances was 31.4% after gynecologic surgery, 31.9% after urologic surgery, and 35.9% after spine surgery. The occurrence of sleep disturbances is associated with worse perioperative outcomes, including aggravated pain intensity, increased delirium, higher risk of cardiovascular events, and delayed hospital discharge.

Dexmedetomidine is a high-specific alpha 2-adrenergic agonist with anxiolytic, sedative, and analgesic effects. When used during general anesthesia and for postoperative analgesia, dexmedetomidine is associated with improved analgesia and sleep quality. The effect of dexmedetomidine is dose-dependent. However, even commonly used dosage increases bradycardia and hypotension.

Ketamine is a non-competitive N-methyl-D-aspartate (NMDA) receptor antagonist. Esketamine is the S-enantiomer of racemic ketamine with a higher affinity for NMDA receptors and is approximately twice as potent as racemic ketamine in analgesia. When used during general anesthesia and for postoperative analgesia, esketamine improves analgesia and reduces opioid consumption, but psychiatric symptoms may occur.

The sedative effect of dexmedetomidine is helpful to relieve psychiatric side effects of ketamine/esketamine. A previous study showed that dexmedetomidine-esketamine combination as a supplement to patient-controlled intravenous analgesia improved postoperative analgesia and subjective sleep quality in patients after scoliosis correction surgery.

This trial is designed to test the hypothesis that dexmedetomidine-esketamine combination used as a supplement during general anesthesia and postoperative intravenous analgesia may reduce sleep disturbances in adult after major noncardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years.
2. Scheduled for major noncardiac surgery (≥60 minutes) under general anesthesia with an expected end of surgery no later than 18:00 pm.
3. Required patient-controlled intravenous analgesia after surgery.

Exclusion Criteria:

1. Emergency surgery, transurethral surgery, organ transplantation.
2. Pregnant or lactating women.
3. Patients who need hypnotics for sleep disturbance or antidepressants for depression prior to surgery.
4. History of schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis.
5. Inability to communicate due to coma, severe dementia, or speech disorders, endured hypoxic encephalopathy or traumatic brain injury, or after neurosurgery.
6. Comorbid with hyperthyroidism and pheochromocytoma.
7. Preoperative left ventricular ejection fraction <30%, sick sinus syndrome, severe sinus bradycardia (heart rate <50 beats/min), atrioventricular block of degree II or higher without pacemaker implantation, or systolic blood pressure below 90 mmHg despite use of vasopressors.
8. Diagnosed as sleep apnea, or judged to be at high risk of moderate-to-severe sleep apnea as assessed by STOP-Bang.
9. Severe hepatic dysfunction (Child-Pugh class C), severe renal dysfunction (on dialysis), or ASA classification ≥IV.
10. Hypersensitive to dexmedetomidine and/or esketamine.
11. Other conditions that are deemed unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of sleep disturbances within 3 days after surgery | Up to 3 days after surgery
  Sleep disturbances are defined as Richards-Campbell Sleep Questionnaire (RCSQ) score below 50, based on assessments conducted daily between 8:00 am and 10:00 am during postoperative days 1 to 3.

SECONDARY OUTCOMES:
Quality of recovery at 24 hours after surgery | At 24 hours after surgery
  Quality of recovery is assessed using the Quality of Recovery-15 (QoR-15) scale at 24 hours after surgery. The total QoR-15 scores are evaluated based on physical comfort (five items), emotional state (four items), psychological support (two items), physical independence (two items), and pain (two items) for QoR-15 questionnaire. Each item is scored from 0 to 10, and the possible total score ranges from 0 to 150, with higher scores representing better recovery quality after operation.
Subjective sleep quality in the first 3 nights after surgery. | Up to 3 days after surgery.
  Subjective sleep quality is assessed daily (8:00 am to 10:00 am) using the Richards-Campbell Sleep Questionnaire (RCSQ) during the first 3 postoperative days. Richards-Campbell Sleep Questionnaire (RCSQ) comprises five items: sleep depth, sleep latency, awakenings, returning to sleep, and sleep quality. Each item is assessed with a 100-mm visual analog scale. The scores range from 0, indicating the worst possible sleep, to 100, indicating the best possible sleep. The total RCSQ sleep score is derived by summing up the individual scores on the five sleep items and dividing it by 5.
Pain intensity both at rest and with movement during the first 3 postoperative days | Up to 3 days after surgery
  Pain intensity is assessed with the numeric rating scale (NRS; an 11-point scale where 0=no pain and 10=the worst pain) twice daily (8:00 am to 10:00 am, and 18:00 pm to 20:00 pm) both at rest and with movement during the first 3 postoperative days.
Anxiety and depression on the third day after surgery | On the third day after surgery
  Postoperative anxiety and depression are assessed using the Hospital Anxiety and Depression Scale (HADS), with scores categorized as follows: 0-7 (negative), 8-10 (mild), 11-14 (moderate), and 15-21 (severe).
Subjective sleep quality on the 30th day after surgery | On the 30th day after surgery
  Subjective sleep quality is assessed with the Pittsburgh Sleep Quality Index (PSQI) on the 30th postoperative day.

OTHER OUTCOMES:
Time to extubation after surgery | On the day of surgery
  Time interval from end of surgery to extubation.
Incidence of emergence agitation after surgery | Up to 2 hours after extubation
  Emergence agitation was defined as a Richmond Agitation-Sedation Scale (RASS) score ≥ +2 at any time point from tracheal extubation to discharge from the post-anesthesia care unit (PACU)
Cumulative opioid consumption within 48 hours after surgery | Within 48 hours after surgery
  Cumulative opioid consumption from end of surgery to 48 hours after surgery.
Proportion of patients requiring rescue analgesia within 48 hours after surgery | Within 48 hours after surgery
  Rescue analgesia indicates any analgesics in addition to patient-controlled intravenous analgesia.
Length of hospital stay after surgery | Up to 30 days after surgery.
  Time interval from end of surgery to hospital discharge.
Agitation and sedation levels during the first 3 postoperative days | Up to 3 days after surgery
  Agitation and sedation levels are assessed using the Richmond Agitation-Sedation Scale (RASS) twice daily (8:00 am to 10:00 am, and 18:00 pm -20:00) during the first 3 postoperative days.
Incidence of postoperative complications | Up to 30 days after surgery
  Postoperative complications are defined as new onset conditions that are deemed harmful and and require therapeutic intervention, i.e., class II or above on the Clavien-Dindo classification.
All-cause 30-day mortality | Up to 30 days after surgery
  All-cause death within 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, Study Chair — Dong-Xin Wang, MD, PhD, Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen RW, Burney CP, Davis A, Henkin J, Kelly J, Judd BG, Ivatury SJ. Deep Sleep and Beeps: Sleep Quality Improvement Project in General Surgery Patients. J Am Coll Surg. 2021 Jun;232(6):882-888. doi: 10.1016/j.jamcollsurg.2021.02.010. Epub 2021 Mar 3. PMID 33675989
- [Background] Myles PS, Shulman MA, Reilly J, Kasza J, Romero L. Measurement of quality of recovery after surgery using the 15-item quality of recovery scale: a systematic review and meta-analysis. Br J Anaesth. 2022 Jun;128(6):1029-1039. doi: 10.1016/j.bja.2022.03.009. Epub 2022 Apr 14. PMID 35430086
- [Background] Kjolhede P, Langstrom P, Nilsson P, Wodlin NB, Nilsson L. The impact of quality of sleep on recovery from fast-track abdominal hysterectomy. J Clin Sleep Med. 2012 Aug 15;8(4):395-402. doi: 10.5664/jcsm.2032. PMID 22893770
- [Background] Gulam S, Xyrichis A, Lee GA. Still too noisy - An audit of sleep quality in trauma and orthopaedic patients. Int Emerg Nurs. 2020 Mar;49:100812. doi: 10.1016/j.ienj.2019.100812. Epub 2020 Jan 30. PMID 32007403
- [Background] Ruiz FS, Andersen ML, Guindalini C, Araujo LP, Lopes JD, Tufik S. Sleep influences the immune response and the rejection process alters sleep pattern: Evidence from a skin allograft model in mice. Brain Behav Immun. 2017 Mar;61:274-288. doi: 10.1016/j.bbi.2016.12.027. Epub 2017 Jan 7. PMID 28069386
- [Background] Chouchou F, Khoury S, Chauny JM, Denis R, Lavigne GJ. Postoperative sleep disruptions: a potential catalyst of acute pain? Sleep Med Rev. 2014 Jun;18(3):273-82. doi: 10.1016/j.smrv.2013.07.002. Epub 2013 Sep 24. PMID 24074687
- [Background] Fernandes NM, Nield LE, Popel N, Cantor WJ, Plante S, Goldman L, Prabhakar M, Manlhiot C, McCrindle BW, Miner SE. Symptoms of disturbed sleep predict major adverse cardiac events after percutaneous coronary intervention. Can J Cardiol. 2014 Jan;30(1):118-24. doi: 10.1016/j.cjca.2013.07.009. Epub 2013 Oct 16. PMID 24140074
- [Background] Lu Y, Li YW, Wang L, Lydic R, Baghdoyan HA, Shi XY, Zhang H. Promoting sleep and circadian health may prevent postoperative delirium: A systematic review and meta-analysis of randomized clinical trials. Sleep Med Rev. 2019 Dec;48:101207. doi: 10.1016/j.smrv.2019.08.001. Epub 2019 Aug 22. PMID 31505369
- [Background] Wang X, Hua D, Tang X, Li S, Sun R, Xie Z, Zhou Z, Zhao Y, Wang J, Li S, Luo A. The Role of Perioperative Sleep Disturbance in Postoperative Neurocognitive Disorders. Nat Sci Sleep. 2021 Aug 6;13:1395-1410. doi: 10.2147/NSS.S320745. eCollection 2021. PMID 34393534
- [Background] Meewisse AJG, Gribnau A, Thiessen SE, Stenvers DJ, Hermanides J, van Zuylen ML. Effect of time of day on outcomes in elective surgery: a systematic review. Anaesthesia. 2024 Dec;79(12):1325-1334. doi: 10.1111/anae.16395. Epub 2024 Aug 7. PMID 39108199
- [Background] Song B, Li Y, Teng X, Li X, Yang Y, Zhu J. Comparison of Morning and Evening Operation Under General Anesthesia on Intraoperative Anesthetic Requirement, Postoperative Sleep Quality, and Pain: A Randomized Controlled Trial. Nat Sci Sleep. 2020 Jul 16;12:467-475. doi: 10.2147/NSS.S257896. eCollection 2020. PMID 32765143
- [Background] Luo M, Song B, Zhu J. Sleep Disturbances After General Anesthesia: Current Perspectives. Front Neurol. 2020 Jul 8;11:629. doi: 10.3389/fneur.2020.00629. eCollection 2020. PMID 32733363
- [Background] Chung F, Liao P, Elsaid H, Shapiro CM, Kang W. Factors associated with postoperative exacerbation of sleep-disordered breathing. Anesthesiology. 2014 Feb;120(2):299-311. doi: 10.1097/ALN.0000000000000041. PMID 24158050
- [Background] Duan G, Wang K, Peng T, Wu Z, Li H. The Effects of Intraoperative Dexmedetomidine Use and Its Different Dose on Postoperative Sleep Disturbance in Patients Who Have Undergone Non-Cardiac Major Surgery: A Real-World Cohort Study. Nat Sci Sleep. 2020 Mar 12;12:209-219. doi: 10.2147/NSS.S239706. eCollection 2020. PMID 32210652
- [Background] Su X, Wang DX. Improve postoperative sleep: what can we do? Curr Opin Anaesthesiol. 2018 Feb;31(1):83-88. doi: 10.1097/ACO.0000000000000538. PMID 29120927
- [Background] Krenk L, Jennum P, Kehlet H. Sleep disturbances after fast-track hip and knee arthroplasty. Br J Anaesth. 2012 Nov;109(5):769-75. doi: 10.1093/bja/aes252. Epub 2012 Jul 24. PMID 22831887
- [Background] Gogenur I, Wildschiotz G, Rosenberg J. Circadian distribution of sleep phases after major abdominal surgery. Br J Anaesth. 2008 Jan;100(1):45-9. doi: 10.1093/bja/aem340. Epub 2007 Nov 23. PMID 18037670